CLINICAL TRIAL: NCT02343315
Title: Effectiveness of TENS and Supervised Motor Control Exercises Compared To Unsupervised Exercises in Subjects With Chronic Low Back Pain: A Randomized Clinical Trial
Brief Title: Are Supervised Exercises and TENS Necessary Along With Prescribed Home Exercises for Chronic Low Back Pain?
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We were unable to run the trial because of inadequate resources (staffing). The principal investigator also moved countries.
Sponsor: Kathmandu University School of Medical Sciences (Other)
Responsible Party: Principal Investigator, Saurab Sharma, MPT, Kathmandu University School of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KUSMS107/14
Record Dates: First submitted 2015-01-15; First posted 2015-01-22 (Estimated); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Chronic Low Back Pain
Keywords: low back pain; home exercises; chronic pain; supervised exercise; core stability exercises; spinal stabilization exercises
MeSH Terms: conditions — Low Back Pain; Chronic Pain | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- TENS (Experimental): Participants will receive Active-TENS along with SMCE and UHEP. Six treatment sessions will be given over two weeks. Total duration of the treatment session may last from 40 - 60 minutes.
  Interventions: Device: TENS; Other: SMCE; Other: UHEP
- SMCE (Experimental): Participants will receive SMCE and UHEP. Six sessions of supervised Motor control exercises will be provided over the period of two weeks.
  Interventions: Other: SMCE; Other: UHEP
- UHEP (Active Comparator): Unsupervised home exercise program will be prescribed with home exercise leaflet and education leaflet in the form of back book on first treatment session.
  Interventions: Other: UHEP

INTERVENTIONS:
Device: TENS — Six treatment sessions will be given over two weeks. Total duration of the treatment session may last from 40 - 60 minutes.
  * Equipment- TENS (CEFAR Basic TENS Machine)
  * Electrodes- Four channel electrode to cover the site of pain
  * Site of electrode placement- will be decided by the physical therapist to best suit or cover the area of pain based on complaints of patient based on the body chart.
  * Intensity- the intensity will be increased progressively until maximum tolerable intensity is reached. This stimulation may cause visible muscle contraction. This type of current is also referred to as Motor-level TENS, which is effective for chronic pain. The intensity will not be increased beyond 25 milli Amperes if no sensation is perceived by the patient.
  * Frequency- 5 Hertz
  * Duration- 30 minutes
  Other Names: transcutaneous electrical nerve stimulation; transcutenous nerve stimulation; transcutaneous electrical stimulation; Low TENS; Motor level TENS
  Arms: TENS
Other: SMCE — Six sessions of supervised Motor control exercises will be provided over the period of two weeks. Exercises will be provided in order to target the function of core muscles of the spine. Each participant in the SMCE group will be trained by a physical therapist to recruit the deep muscles of the spine and reduce the activity of superficial muscles.
  Initially participants will be taught how to contract the transversus abdominis and multiﬁdus muscles in isolation from the more superﬁcial trunk muscles, but in conjunction with the pelvic ﬂoor muscles. Pressure biofeedback will be used in order to provide feedback about muscle recruitment to the participant. Exercises will be provided to the participants in the progressive manner. Later, movement of limbs will be incorporated with the contraction of the core muscles. Finally, these core muscle activation will be emphasized during the functional activities.
  Other Names: core stability exercises; spinal stabilization exercises; Supervised motor control exercises
  Arms: SMCE; TENS
Other: UHEP — All the participants will receive the following treatments:
  1. Unsupervised home exercise program- which includes series of motor control exercises along with specific exercises including stretching exercises based on impairments.
  2. Education in terms of body mechanics, ergonomics advises and educational leaflet in the form of Nepali version of Back book which includes, evidence based advises about back pain self-management, advice to remain active. Treating physical therapist will educate all the participants in the first intervention session.
  3. Participants will not be asked to not take the "over the counter" analgesics including Acetaminophen or Non-inflammatory anti-inflammatory drugs (ibuprofen).
  Other Names: home exercise program; Unsupervised home exercise program

SUMMARY:
The purpose of this study is to compare the added effects of TENS and Supervised Motor Control Exercises (SMCE) over Unsupervised Home Exercise Program (UHEP) on disability, pain and other outcomes.

DETAILED DESCRIPTION:
Chronic low back pain (CLBP) is a common problem causing disability and high economic burden in globally as well as in Nepal. There is no consensus on treatment of CLBP, however motor control exercises have good evidence on improvement in pain and disability in CLBP population, whereas transcutaneous electrical nerve stimulation (TENS) is a common treatment of choice with some evidence. But, we do not know if supervising these motor control exercises (SMCE) and TENS have any added benefit over home exercise program (HEP) which is commonly prescribed mode of exercises. We plan to conduct a three armed randomized control trial to answer this question to compare effects of SMCE, TENS and HEP versus SMCE and HEP versus HEP alone on disability and pain at two weeks and six months follow up. Three way-mixed model analysis of Variance (ANOVA) will be used as the statistical test. Appropriate post hoc analysis will be done to compare within group and between group differences.

ELIGIBILITY:
Inclusion Criteria:

1. Nonspecific Low back pain for more than 3 months with pain primarily localized between T12 and gluteal folds, if patients report that their pain is provoked and relieved with postures, movement and activities.
2. Age between 18 to 65 years
3. Male or female
4. All educational backgrounds (educated or uneducated)
5. Pain intensity more than 2/10 on NPRS and
6. Disability of more than 20/100 on NODI

Exclusion Criteria:

1. Red flags noted in the participant's general medical screening questionnaire (i.e. tumor, metabolic diseases, Rheumatoid Arthritis, osteoporosis, prolonged history of steroid use, etc.)
2. Signs consistent with nerve root compression, this includes any one of the following:

   1. Reproduction of low back or leg pain with straight leg raise at less than 45 degrees
   2. Muscle weakness involving a major muscle group of the lower extremity
   3. Diminished lower extremity muscle stretch reflex (Quadriceps or Achilles tendon)
   4. Diminished or absent sensation to pinprick in any lower extremity dermatome
3. Prior surgery to the lumbar spine or buttock
4. Current pregnancy
5. Past medical history of osteoporosis or spinal compression fracture
6. Participants who do not provide informed consent for the study

   -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-08 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Disability (Nepali version of Oswestry Disability Index (NODI) | 2 weeks
  Nepali version of Oswestry Disability Index (NODI) will be used to measure disability which is a cross culturally adapted and validated tool for measuring disability in low back pain population in Nepal. The tool has acceptable reliability (Cronbach's Alpha= 0.723, intraclass correlation coefficient= 0.875)

SECONDARY OUTCOMES:
Pain intensity (Numerical Pain Rating Scale (NPRS) | 2 weeks
  Numerical Pain Rating Scale (NPRS) - An 11-point numeric pain rating scale ranging from 0 (no pain) to 10 (worst imaginable pain) will be used to assess current pain intensity and the best and worst level of pain during the last 24 hours.
Pain intensity (Numerical Pain Rating Scale (NPRS) | 6 months
  Numerical Pain Rating Scale (NPRS) - An 11-point numeric pain rating scale ranging from 0 (no pain) to 10 (worst imaginable pain) will be used to assess current pain intensity and the best and worst level of pain during the last 24 hours.
Disability (Nepali version of Oswestry Disability Index (NODI) | 6 months
  Nepali version of Oswestry Disability Index (NODI) will be used to measure disability which is a cross culturally adapted and validated tool for measuring disability in low back pain population in Nepal. The tool has acceptable reliability (Cronbach's Alpha= 0.723, intraclass correlation coefficient= 0.875)

OTHER OUTCOMES:
Changes in pain and disability (Global Rating of Change (GROC) | 2 weeks
  Global Rating of Change (GROC) - The fifteen-point global rating scale will be used. The scale ranges from -7 (a very great deal worse) to zero (about the same) to +7 (a very great deal better). Intermittent descriptors of worsening or improving are assigned values from -1 to -6 and +1 to +6 respectively. The global rating will be administered at the follow-up examinations only.
Changes in pain and disability (Global Rating of Change (GROC) | 6 months
  Using Global rating of change (GROC)
Need for medication (using frequency and dosage and types of analgesics used) | 6 months
  using frequency and dosage and types of analgesics used
Need for follow up (number of treatment sessions in past six months will be recorded) | 6 months
  number of treatment sessions in past six months will be recorded
Adverse events | 6 months
  numbers of adverse events are noted down using a questionnaire
Fear avoidance (Fear avoidance belief questionnaire (FABQ) | 6 months
  Fear avoidance belief questionnaire (FABQ) - The FABQ is a 16-item scale that assesses the influence of fear avoidance behaviors on physical and work activities. Each item is scored from 0-6 with possible scores ranging between 0-42 and higher scores representing increased fear-avoidance beliefs.
Pain Catastrophizing (Pain catastrophizing Scale (PCS) | 6 months
  Pain catastrophizing Scale (PCS) - Nepali translation of PCS is a 13-item scale that assesses the pain catastrophizing. Pain catastrophizing is an exaggerated, negative focus on pain and is related to psychological distress, pain severity, and other negative outcomes in pain population. Participants responded to each item using a Likert-type scale from 0 ('not at all') to 4 ('all the time').

CONTACTS AND LOCATIONS:
Overall Officials: Saurab Sharma, MPT, Principal Investigator — Kathmandu University School of Medical Sciences, Nepal